CLINICAL TRIAL: NCT01387360
Title: A Prospective Study to Evaluate the Safety and Effectiveness of the Supracor Presbyopic Treatment Algorithm for Pseudophakic Eyes Using Lasik
Brief Title: Presbyopic Supracor Treatment for Near Myopic/Hyperopic Pseudophakic Eyes
Acronym: SUPRACOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1107
Record Dates: First submitted 2011-06-28; First posted 2011-07-04 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Myopia; Hyperopia; Presbyopia
Keywords: Myopia; Hyperopia; Presbyopia; Pseudophakia; LASIK
MeSH Terms: conditions — Myopia; Hyperopia; Presbyopia; Pseudophakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supracor (Experimental): Study arm will consist of patients who have undergone previous cataract surgery with implantation of a monofocal IOL. The Supracor procedure will be performed on the non-dominant pseudophakic eye of these patients.
  Interventions: Device: Supracor

INTERVENTIONS:
Device: Supracor — The presbyopic treatment consists of a standard treatment for distance vision and the procedure known as SUPRACOR addition to correct near vision.
  The SUPRACOR addition provides a multifocal ablation with a central near addition with an aberration controlled transition zone towards the periphery, thereby allowing good focus over a range of object distances.
  Other Names: PresbyLASIK; Multifocal Ablation

SUMMARY:
This clinical study has been planned to determine the effectiveness of a special laser treatment intended to correct both near and distance vision in patients who have undergone previous cataract surgery.

DETAILED DESCRIPTION:
This clinical study has been planned to evaluate the safety and effectiveness of the SUPRACOR presbyopic excimer laser treatment algorithm for near myopic and near hyperopic indications, with or without astigmatism, when performed on the cornea of pseudophakic eyes implanted with a monofocal IOL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 45 years old
* Subjects must read, understand, and sign an Informed Consent Form (ICF).
* Subjects must be willing and able to return for scheduled follow-up examinations through 6 months after surgery.
* Subjects must have undergone previous uncomplicated cataract surgery with monofocal IOL implant in the study eye at least 3 months prior to study enrollment.
* Subjects must have up to +/- 2.0 (D) of absolute spherical myopia or hyperopia (not spherical equivalent), with up to +/- 2.0 D of refractive astigmatism (NOT corneal astigmatism) by manifest subjective refraction. The spherical equivalent must be no more than +/- 2.0 D.
* Subjects who have be screened successfully for acceptance of the SUPRACOR simulation

Exclusion Criteria:

* Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining corneal thickness below the flap postoperatively.
* Subjects for whom the preoperative assessment of the ocular topography indicates that one or both eyes are not suitable candidates for treatment based upon the suggested computer-simulated treatment plan (e.G. Keratoconus).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The percentage of treated eyes with a best corrected high contrast distance VA of 20/25 or better | 6M

SECONDARY OUTCOMES:
The percentage of treated eyes within +/- 1.00D of target refraction | 6M
The percentage of treated eyes within +/- 0.50D of target refraction | 6M
The percentage of treated eyes with an uncorrected high contrast near VA of 20/40 or better | 6M
Stability analysis: change of ≤ 1D MRSE between two consecutive post-op visits | 6M
Preservation of VA: Loss of more than 2 lines in BCVA for distance vision | 6M
The percentage of treated eyes with a best-distance corrected high contrast distance VA of 20/40 or better | 6M
The percentage of treated eyes with an induced subjective manifest refraction cylinder not within +/- 2.00D | 6M
Cumulative incidence of AEs | 6M
Cumulative incidence subjective symptoms | 6M

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ang, M.D., Study Director — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati, Manila, Philippines

REFERENCES:
- [Background] Pinelli R. More on peripheral PresbyLASIK as a center-distance technique. J Refract Surg. 2008 Sep;24(7):665. doi: 10.3928/1081597X-20080901-04. No abstract available. PMID 18811107
- [Background] de Ortueta D. Is peripheral presbyLASIK a center-distance technique? J Refract Surg. 2008 Jun;24(6):561; author reply 562. doi: 10.3928/1081597X-20080601-01. No abstract available. PMID 18581778
- [Result] Epstein RL, Gurgos MA. Presbyopia treatment by monocular peripheral presbyLASIK. J Refract Surg. 2009 Jun;25(6):516-23. doi: 10.3928/1081597X-20090512-05. PMID 19603619
- [Result] Alio JL, Amparo F, Ortiz D, Moreno L. Corneal multifocality with excimer laser for presbyopia correction. Curr Opin Ophthalmol. 2009 Jul;20(4):264-71. doi: 10.1097/icu.0b013e32832a7ded. PMID 19537363
- [Result] Pinelli R, Ortiz D, Simonetto A, Bacchi C, Sala E, Alio JL. Correction of presbyopia in hyperopia with a center-distance, paracentral-near technique using the Technolas 217z platform. J Refract Surg. 2008 May;24(5):494-500. doi: 10.3928/1081597X-20080501-07. PMID 18494342
- [Result] Ortiz D, Alio JL, Illueca C, Mas D, Sala E, Perez J, Espinosa J. Optical analysis of presbyLASIK treatment by a light propagation algorithm. J Refract Surg. 2007 Jan;23(1):39-44. doi: 10.3928/1081-597X-20070101-07. PMID 17269242